CLINICAL TRIAL: NCT06250010
Title: Immunotolerance in Endometrial Cancer and at the Maternal-fetal Interface: Immunological
Brief Title: Immunotolerance in Endometrial Cancer and at the Maternal-fetal Interface: Immunological Profiling of the Tumor Microenvironment in Risk Stratification of Recurrence
Status: Recruiting | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: Federico II University (Other)
Responsible Party: Sponsor
Other Study IDs: RS1807/22
Record Dates: First submitted 2024-01-16; First posted 2024-02-08 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Endometrial tissue samples taken from surgically treated patients and samples of decidualized endometrium and trophoblast from patients with ongoing spontaneous abortion treated surgically
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: tissue samples (healthy and tumor taken from the same patient): Tissue samples (healthy and tumor taken from the same patient) collected at the Institute's Biobank (starting from 2017) (retro-prospective). The data relating to the neoplastic pathology will also be indicated: histotype, grading, FIGO stage. And data on oncological follow-up: any intra or post-operative complications, any adjuvant therapies, type and date of any recurrence/metastasis, type of treatment, any recurrence, date and manner of death
  Interventions: Diagnostic Test: tissue samples (healthy and tumor taken from the same patient) and tissue samples (decidualized endometrium and trophoblast taken from it patient)
- Cohort 2: tissue samples (decidualized endometrium and trophoblast taken from it patient): The tissue samples (decidualized endometrium and trophoblast taken from it patient) which will be collected from the Gynecology and Obstetrics Unit of the Polyclinic Federico II University of Naples (prospective) and transferred to the Regina National Cancer Institute Elena, IRE-IFO
  Interventions: Diagnostic Test: tissue samples (healthy and tumor taken from the same patient) and tissue samples (decidualized endometrium and trophoblast taken from it patient)

INTERVENTIONS:
Diagnostic Test: tissue samples (healthy and tumor taken from the same patient) and tissue samples (decidualized endometrium and trophoblast taken from it patient) — Correlation between the immuno-score results of each patient with his prognosis, in terms disease-free survival, overall survival, relapse-free survival, disease-specific survival cancer, distant and/or local free survival, to validate their potential role independent in the progression of endometrial cancer; later, for a better characterization of the various ones risk classes, we will combine our immuno-score with the already known risk factors, included in the ESMO-ESGO-ESTRO classification and in the biomolecular classification of endometrial cancer, to investigate whether the Microenvironmental immunological factors in endometrial cancer could allow better stratification of patients in risk classes.

SUMMARY:
This pilot/exploratory study will be configured as a non-retro-prospective study interventional on endometrial tissue samples taken from surgically treated patients at the Regina Elena National Cancer Institute, IRE - IFO and stored at the Biobank of same Institute (BBIRE) (cohort 1) and on samples of decidualized endometrium and trophoblast from patients with ongoing spontaneous abortion treated surgically at the UOC of Gynecology ed Obstetrics of the Federico II University Polyclinic of Naples (cohort 2)

DETAILED DESCRIPTION:
For the experiments proposed in the project the following will be used:

Court 1: tissue samples (healthy and tumor taken from the same patient) collected at the Institute's Biobank (starting from 2017) (retro-prospective); Court 2: tissue samples (decidualized endometrium and trophoblast taken from it patient) which will be collected at the Gynecology and Obstetrics Unit of the Polyclinic Federico II University of Naples (prospective) and transfer to the Regina National Cancer Institute Elena, IRE-IFO.

Clinical data

The following data will be collected for each patient:

* Age, ethnicity, parity, luxury habits, level of education, marital status, height, weight, index of body mass
* Data on previous clinical history, previous gynecological-obstetric pathologies and any treatments, current comorbidities and medical therapies

For Cohort1 patients only:

* Data relating to the neoplastic pathology: histotype, grading, FIGO stage
* Data on oncological follow-up: any intra- or post-operative complications, any therapies adjuvants, type and data of any recurrence/metastasis, type of treatment if any recurrence, date and manner of death.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1: Oncology patients

* Age >18 years
* Histological diagnosis of endometrial hyperplasia with and without atypia, endometrial carcinoma endometrioid histotype at any stage of the disease (FIGO I-IV), patients subjected to hysterectomy for benign extra-endometrial pathology, patients with recurrence/metastasis from endometrioid endometrial carcinoma who undergo surgery;
* Adequate biological material to be able to carry out the planned analyses;
* Written informed consent (only for patients in the prospective part and/or in follow up/traceable);
* For the retrospective part: availability of samples adequately stored at the biobank of the Institute and availability of data relating to follow-up (at least 36 months).

Cohort 2: Patients with ongoing spontaneous abortion

* Age >18 years;
* Diagnosis of ongoing spontaneous abortion which is subjected to an instrumental review procedure of the uterine cavity, under hysteroscopic guidance;
* Adequate biological material to be able to carry out the analyzes previously described;
* Written informed consent.

Exclusion Criteria:

* Comorbidities not controlled with adequate medical therapy;
* Infections of the endometrial cavity (pyometra);
* Synchronous tumors;
* Neoadjuvant treatments;
* Previous radiation treatments on the pelvic region.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oncology patients who have undergone or will undergo to surgery. And patients with ongoing miscarriage who do will undergo surgery.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-12-13 (Actual); Primary Completion 2025-12-13 (Estimated); Study Completion 2025-12-13 (Estimated)

PRIMARY OUTCOMES:
Description of genetic signatures shared between the maternal-fetal interface | 36 months
  The trial aims to describe gene signatures shared between the maternal-fetal interface and the various stages of progression of endometrial carcinoma, through transcriptomic analysis, with the aim of evaluate their functional role in the immune escape of endometrial carcinoma.Transcriptomics (RNA-seq) coupled with will be used imaging approaches (IHC) and digital pathology. Spatial techniques will be exploited transcriptomics coupled to single-cell RNA-seq to study interactions between cells in the TME and at the maternal-fetal interface. The results of each patient's immuno-score will be correlated with his prognosis, in terms disease-free survival, overall survival, relapse-free survival, disease-specific survival cancer, distant and/or local free survival, to validate their potential role independent in the progression of endometrial cancer.
Calculation of potential immuno-score | 36 months
  Calculation of potential immuno-score for each patient, considering immune pathways, correlating the results of each patient's immuno-score with his prognosis, in terms disease-free survival and overall survival.
characterize the risk classes | 36 months
  To characterize the various risk classes, the immuno-score will be combined with the already known risk factors, included in the ESMO-ESGO-ESTRO classification and in the biomolecular classification of endometrial carcinoma, to investigate whether the Microenvironmental immunological factors in endometrial cancer might allow for better stratification of patients in risk classes, with the use of Artificial Intelligence, such as Machine Learning and neural networks.

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Bruno, Doctor, Principal Investigator — IRCCS "Regina Elena" National Cancer Institute
Locations (1):
- "Regina Elena" National Cancer Institute, Rome, Italy